CLINICAL TRIAL: NCT01852474
Title: Effects of tDCS in Cortical Plasticity and Motor Learning in Children With Cerebral Palsy
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Motor Learning in Children With Cerebral Palsy (CP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Pedal with Pete (Unknown)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-p-000629
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Palsy
Keywords: motor learning; cortical plasticity; direct current stimulation
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active tDCS (Experimental): Subjects will receive active tDCS stimulation for 5 sessions (20m/each) over one week.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Subjects will receive tDCS stimulation 1x per day for 5 days (over the period of 1 week). Each session will be 20 minutes long. The subject will receive active stimulation for the entire 20 minutes.
  Other Names: 1x1 direct current stimulator; soterix medical; transcranial stimulation

SUMMARY:
In this study, the investigators aim to assess the clinical and neurophysiological effects of a non-invasive brain stimulation technique - transcranial direct current stimulation (tDCS)- on cortical plasticity and motor learning in children with cerebral palsy. Investigators will use different assessment techniques, such as transcranial magnetic stimulation (TMS) and kinematics (sensors) to measure changes through the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants must be between 8 and 18 years old.
* Diagnosis of spastic or mixed CP with distribution of diplegia and/or hemiplegia form.
* Gross Motor Function Classification System for Cerebral Palsy (GMFCS) level II and III.
* Manual Ability Classification System for Children with CP (MACS) level II up to IV.
* Ability to cooperate and follow directions.

Exclusion Criteria:

* Muscle tone reduction therapy in the past 3 months prior to study onset.
* Upper limb orthopedic surgery in the past 3 months prior to study onset.
* Any other form of therapy or procedure involving motor neuron junction inhibition; either by biochemical and/or mechanical denervation, in the past 3 months prior to study onset.
* History of convulsive disorder in the past 2 years prior to study onset.
* Current use of carbamazepine as anticonvulsive therapy.
* Presence ventriculoperitoneal shunt.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in motor assessments | Approximately 2 weeks
  Investigators will measure changes in kinematic (sensor) assessments from baseline to follow-up. The sensor will collect Inertial Measurements Units (IMU) and complex motion sensing, as measured by accelerometer/gyroscope/magnetometer of freedom motion capture.

SECONDARY OUTCOMES:
Changes in TMS measurements | Approximately 2 weeks
  Investigators will measure change in TMS measurements from baseline to follow-up. TMS measures will consist of: motor threshold, motor evoked potentials (MEP's), transcallosal inhibition, and examinations of intracortical inhibition and facilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States